CLINICAL TRIAL: NCT00432159
Title: A Multi-Center, Prospective, Randomized Controlled Trial Comparing Cervical Arthroplasty to Anterior Cervical Discectomy and Fusion for the Treatment of Cervical Degenerative Disc Disease
Brief Title: Comparison of DISCOVER™ Artificial Cervical Disc and ACDF for Treatment of Cervical DDD (IDE Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DePuy Spine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-DISCOVER
Record Dates: First submitted 2007-02-05; First posted 2007-02-07 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-09

CONDITIONS: Cervical Degenerative Disc Disease
Keywords: cervical; spinal; arthroplasty; disc; surgical; ACDF; DDD
MeSH Terms: interventions — Bone Plates

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participant was masked to which treatment they would receive until AFTER the surgery/treatment procedure. At that point, they were unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- 1-level Cervical TDR (Experimental): Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at a single level of the cervical spine, C3 to C7 inclusive.
  Interventions: Device: Cervical TDR
- 1-level ACDF with plate (Active Comparator): Anterior Cervical Discectomy and Fusion with plate (ACDF with plate) using allograft spacer and the SLIM-LOC™ Anterior Cervical Plate System at a single level of the cervical spine, C3 to C7 inclusive.
  Interventions: Device: ACDF with plate
- 2-level Cervical TDR (Experimental): Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at two adjacent levels of the cervical spine, C3 to C7 inclusive.
  Interventions: Device: Cervical TDR
- 2-level ACDF (Active Comparator): Anterior Cervical Discectomy and Fusion with plate (ACDF with plate) using allograft spacer and the SLIM-LOC™ Anterior Cervical Plate System at two adjacent levels of the cervical spine, C3 to C7 inclusive.
  Interventions: Device: ACDF with plate
- Training: 1 & 2-level Cervical TDR (Experimental): Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at a single level or multiple levels of the cervical spine, C3 to C7 inclusive. Training cohort.
  Interventions: Device: Cervical TDR

INTERVENTIONS:
Device: Cervical TDR — Cervical total disc replacement using a DISCOVER Artificial Cervical Disc.
  Other Names: cervical arthroplasty; cervical disc; c-TDR; DISCOVER disc
  Arms: 1-level Cervical TDR; 2-level Cervical TDR; Training: 1 & 2-level Cervical TDR
Device: ACDF with plate — Anterior cervical discectomy followed by insertion of allograft spacer and placement of an anterior plate.
  Other Names: ACDF; Slim-Loc; Anterior cervical discectomy and fusion with plate
  Arms: 1-level ACDF with plate; 2-level ACDF

SUMMARY:
This study is intended to treat patients with symptomatic degenerative disc disease at one level of the cervical spine. The patients will be randomized to the DISCOVER Artificial Cervical Disc (total disc replacement) or SLIM-LOC™ (cervical fusion) to determine the safety and efficacy at 2 years post operative. Follow-up on patients treated with total disc replacement will be continued to 5 years post operative.

DETAILED DESCRIPTION:
This study is designed as a multicenter, prospective, randomized, controlled trial. Subjects will be stratified by the number of levels to be treated then assigned treatment in a randomized 1:1 ratio. Participants in the treatment group will undergo cervical total disc replacement with the DISCOVER Artificial Cervical Disc. Participants in the control group will undergo anterior cervical discectomy and fusion with the SLIM-LOC™ Anterior Cervical Plate System with a cortical or cortico-cancellous allograft spacer. Follow-up visits will occur at 2 weeks, 3 and 6 months and 1, and 2 years for all randomized subjects. Subjects that received the control treatment will complete their required study participation at 2 years post operative and subjects assigned the Discover treatment will complete their participation at 5 years post operative. Follow-up for the Discover treatment group will be via a telephone administered questionnaire at 3, 4 and 5 years post operative.

ELIGIBILITY:
Key Inclusion Criteria:

* Objective evidence of cervical disc disease in 1 vertebral level between C3-C7 defined as (a) shoulder and/or arm pain in a documented radicular distribution resulting from herniated disc or bony osteophytes or (b)myeloradiculopathy resulting from mild spinal cord compression and nerve root impingement
* Unresponsiveness to documented non-surgical management for greater than or equal to 6 weeks and/or presentation with progressive symptoms of nerve root or spinal cord compression in the face of continued non-surgical management
* Moderate Neck Disability Index (NDI) score
* Able to give informed consent for study participation
* Able and willing to return for all follow-up visits

Key Exclusion Criteria:

* Significant cervical degenerative disc disease
* Prior fusion procedure at any level(s) (C1-T1)
* Marked cervical instability on lateral or flexion/extension radiographs
* Presence of systemic infection or infection at the surgical site
* Diagnosis of a condition, or requires postoperative medication(s), which may interfere with bony/soft tissue healing
* History of alcohol and/or drug abuse
* Any known allergy to a metal alloy or polyethylene
* Morbid obesity
* Any significant general illness (e.g., metastatic cancer, HIV)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2016-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (30):
  - Olympia Medical Center, Beverly Hills, California
  - Sutter Medical Center, Sacramento, California
  - Rocky Mountain Associates in Orthopedic Medicine, PC, Loveland, Colorado
  - Yale University, New Haven, Connecticut
  - Florida Orthopaedic Institute, Tampa, Florida
  - Emory Orthopaedics and Spine Center, Atlanta, Georgia
  - Rush University/Midwest Orthopaedics, Chicago, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Johnson County Spine, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Boston Spine Group, Newton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Twin Cities Spine, Minneapolis, Minnesota
  - St. John's Regional Medical Center, Springfield, Missouri
  - St. Patrick Hospital Neurological Associates, Missoula, Montana
  - Nebraska Spine Center, LLC, Omaha, Nebraska
  - Center for Diseases and Surgery of the Spine, Las Vegas, Nevada
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Southern NY Neurosurgical Group, Johnson City, New York
  - Upstate Medical College/SUNY, Syracuse, New York
  - Carolina Neurosurgery & Spine Associates, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - Neurospine Institute, Eugene, Oregon
  - North Texas Spine Care at Baylor Health, Dallas, Texas
  - Texas Back Institute, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- Pacific Private Clinic, Queensland, Australia
- St. Elisabeth Ziekenhuis, Tilburg, Netherlands

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on July 10, 2006. The final study subjects were enrolled on March 22, 2011 and all study sites were informed that enrollment was closed effective March 31, 2011.
Groups:
- 1-level Cervical TDR: Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at a single level of the cervical spine, C3 to C7 inclusive. Cervical TDR: Cervical total disc replacement using a DISCOVER Artificial Cervical Disc.
- 1-level ACDF With Plate: Anterior Cervical Discectomy and Fusion with plate (ACDF with plate) using allograft spacer and the SLIM-LOC™ Anterior Cervical Plate System at a single level of the cervical spine, C3 to C7 inclusive. ACDF with plate: Anterior cervical discectomy followed by insertion of allograft spacer and placement of an anterior plate.
- 2-level Cervical TDR: Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at two adjacent levels of the cervical spine, C3 to C7 inclusive. Cervical TDR: Cervical total disc replacement using a DISCOVER Artificial Cervical Disc.
- 2-level ACDF: Anterior Cervical Discectomy and Fusion with plate (ACDF with plate) using allograft spacer and the SLIM-LOC™ Anterior Cervical Plate System at two adjacent levels of the cervical spine, C3 to C7 inclusive. ACDF with plate: Anterior cervical discectomy followed by insertion of allograft spacer and placement of an anterior plate.
- Training: 1 & 2-level Cervical TDR: Cervical Total Disc Replacement (Cervical TDR) arthroplasty with the DISCOVER™ Artificial Cervical Disc at a single or multiple levels of the cervical spine, C3 to C7 inclusive. Training cohort. Cervical TDR: Cervical total disc replacement using a DISCOVER Artificial Cervical Disc.
Period: Overall Study
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Started | 185 | 167 | 39 | 20 | 89
Completed | 163 (Actual (Complete efficacy)) | 137 (Actual (Complete efficacy)) | 35 (Actual (Complete efficacy)) | 15 (Actual (Complete efficacy)) | 79 (Actual (Complete efficacy))
Not Completed | 22 | 30 | 4 | 5 | 10
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Failure | 9 | 5 | 3 | 2 | 3
Not completed — Missing NDI and/or neuro. assessment | 13 | 24 | 1 | 3 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR | Total
Number analyzed (Participants) | 185 | 167 | 39 | 20 | 89 | 500
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (8.63) | 42.8 (7.63) | 44.1 (7.94) | 44.4 (7.74) | 42.3 (7.49) | 43.4 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 89 | 26 | 10 | 42 | 260
  Male | 92 | 78 | 13 | 10 | 47 | 240
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 1 | 1 | 1 | 14
  Not Hispanic or Latino | 172 | 153 | 38 | 19 | 88 | 470
  Unknown or Not Reported | 6 | 10 | 0 | 0 | 0 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 1 | 2 | 1 | 0 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 1 | 2 | 4 | 21
  White | 170 | 147 | 36 | 18 | 82 | 453
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 6 | 11 | 1 | 0 | 0 | 18
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index in units of kilogram per meter squared
  kg/m^2 | 28.3 (4.97) | 27.6 (4.83) | 28.3 (4.97) | 30.0 (3.61) | 28.9 (5.12) | 28.3 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: Subject must show 15 point improvement in the Neck Disability Index from baseline to 24 months post operative as well as have no device related SAE, Secondary Surgical Interventions at the index level or any new permanent neurological deterioration.
Time Frame: 24 months
Population: The primary outcome was analyzed with an Intent to Treat (As Randomized) analysis. The difference between the number of treated patients and the number of participants analyzed for each group at the 24 month visit is due to: death of one randomized ACDF patient and patients with no data for NDI and Neurological function (missing data).
Measure: Number; unit: participants who are successes
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 169 | 133 | 38 | 17 | 82
participants who are successes | 137 | 110 | 28 | 13 | 65

2. Secondary Outcome: NDI Success
Description: 15 point improvement in NDI. NDI has a max score of 50, which is calculated based on the 6 answers to each of the 10 questions. Each answer within a question is given a numerical value 0 to 5.
Time Frame: 24 months
Population: Intent to Treat (As Randomized). The difference between the number of treated patients and the number of participants analyzed is due to: death of one randomized ACDF patient, patients who experienced a Device Failure before the 24 month visit, and patients with no data collected for this secondary outcome (missing data).
Measure: Number; unit: participants who are successes
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 161 | 127 | 35 | 15 | 78
participants who are successes | 139 | 111 | 29 | 13 | 67

3. Secondary Outcome: Neurological Component of Success
Description: no new clinically significant permanent abnormalities in neurological function
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants who are successes
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 162 | 129 | 35 | 15 | 80
participants who are successes | 161 | 127 | 35 | 15 | 77

4. Secondary Outcome: Subsequent Secondary Surgery Component of Success
Description: no subsequent secondary surgical intervention at the index level
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants who are successes
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 185 | 167 | 39 | 20 | 89
participants who are successes | 176 | 160 | 35 | 18 | 84

5. Secondary Outcome: Device-Related SAE Component of Success
Description: no device related serious adverse events
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants who are successes
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 185 | 167 | 39 | 20 | 89
participants who are successes | 184 | 167 | 39 | 20 | 89

6. Secondary Outcome: NDI - Change From Baseline
Description: Change from baseline of the Neck Disability Index. NDI has a minimum score of 0 (no disability) and a maximum score of 50 (complete disability) , which is calculated based on the 6 answers to each of the 10 questions. Each answer within a question is given a numerical value 0 to 5.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: NDI Score
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 161 | 127 | 35 | 15 | 78
NDI Score | -33.4 (17.97) | -33.2 (18.04) | -32.8 (20.62) | -32.9 (22.10) | -34.3 (21.00)

7. Secondary Outcome: Neck Pain VAS Scores - Change From Baseline
Description: Change from baseline of the Neck Pain VAS Scores. VAS is a 100-mm visual analog scale used to assess pain. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their neck.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 124 | 35 | 15 | 78
Units on a scale | -47.0 (30.43) | -41.5 (30.57) | -36.1 (33.15) | -27.2 (26.14) | -46.3 (33.60)

8. Secondary Outcome: Maximum Arm Pain VAS - Change From Baseline
Description: Change from baseline in maximum value of the left and right arm VAS scores. VAS is a 100-mm visual analog scale used to assess pain. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their arm.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 123 | 35 | 15 | 78
Units on a scale | -52.0 (32.69) | -49.5 (33.45) | -42.4 (37.54) | -30.9 (44.62) | -44.3 (35.61)

9. Secondary Outcome: Average Arm Pain VAS - Change From Baseline
Description: Change from baseline in average of the left and right arm VAS scores. VAS is a 100-mm visual analog scale used to assess pain. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their arm.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 123 | 35 | 15 | 78
Units on a scale | -32.1 (25.62) | -28.8 (20.88) | -30.5 (25.90) | -20.6 (26.33) | -26.6 (24.70)

10. Secondary Outcome: Maximum Shoulder Pain VAS - Change From Baseline
Description: Change from baseline in Maximum value of the left and right shoulder VAS scores. VAS is a 100-mm visual analog scale used to assess pain. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their shoulder.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 123 | 35 | 15 | 78
Units on a scale | -52.1 (31.96) | -47.9 (30.18) | -43.0 (34.74) | -21.4 (43.84) | -45.9 (38.13)

11. Secondary Outcome: Average Shoulder Pain VAS - Change From Baseline
Description: Change from baseline in Average of the left and right shoulder VAS scores. VAS is a 100-mm visual analog scale used to assess pain. It asks the subject to place a vertical mark on a 100-mm horizontal line, with 'No pain' listed on the left (at 0 mm) and 'Very severe pain' labeled on the right (at 100 mm). The subject is instructed to indicate the amount of pain they feel in their shoulder.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 123 | 35 | 15 | 78
Units on a scale | -34.1 (26.45) | -31.6 (22.69) | -31.7 (30.36) | -15.6 (24.85) | -31.0 (29.12)

12. Secondary Outcome: Dysphagia Disability Index - Change From Baseline
Description: Change from baseline in Dysphagia Disability Index (DDI). The DDI is designed to evaluate dysphagia, difficulty in swallowing, using a 25-item questionnaire. Responses from the questionnaire were scored as "always" 4, "sometimes" 2, or "never" 0, and summed to provide a total score (range 0-100). Higher DDI scores suggest greater subjective signs of dysphagia.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 154 | 117 | 35 | 15 | 77
Units on a scale | -1.3 (7.91) | 0.7 (7.22) | 0.3 (10.19) | 1.2 (5.89) | -0.8 (9.56)

13. Secondary Outcome: SF-36 - Physical Composite Scores (PCS) - Change From Baseline
Description: Change from baseline in Quality of Life - Physical Composite Scores. SF-36 is based on units on a scale; where 0 is severe disability and 100 is no disability. The scores are scaled (based on weighted sum of the questions)
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 160 | 127 | 35 | 15 | 79
Units on a scale | 14.2 (10.66) | 13.3 (10.50) | 15.2 (9.23) | 6.6 (10.18) | 15.2 (10.73)

14. Secondary Outcome: SF-36 - Mental Composite Scores (MCS) - Change From Baseline
Description: Change from baseline in Quality of Life - Mental Composite Scores. SF-36 is based on units on a scale; where 0 is severe disability and 100 is no disability. The scores are scaled (based on weighted sum of the questions)
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 160 | 127 | 35 | 15 | 79
Units on a scale | 9.2 (11.66) | 8.8 (12.01) | 6.3 (12.89) | 12.2 (13.65) | 6.3 (13.19)

15. Secondary Outcome: Work Status Assessment
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 167 | 131 | 38 | 16 | 83
participants
  Not Working | 28 | 18 | 6 | 2 | 11
  Full Time | 111 | 91 | 21 | 12 | 61
  Part Time | 12 | 10 | 2 | 2 | 7
  Full or Part Time | 123 | 101 | 23 | 14 | 68
  Total | 151 | 119 | 29 | 16 | 79
  Not Applicable | 16 | 12 | 9 | 0 | 4

16. Secondary Outcome: Return to Work
Description: Estimated Proportion of Subjects Returning to Work
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: % of subjects who returned to work
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 172 | 157 | 31 | 20 | 85
% of subjects who returned to work | 87 | 86 | 84 | 90 | 92

17. Secondary Outcome: Activity
Description: Clinical Assessment of Activity
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 162 | 129 | 35 | 15 | 80
participants
  Light | 39 | 30 | 11 | 5 | 21
  Moderate | 79 | 58 | 17 | 8 | 37
  Vigorous | 44 | 41 | 7 | 2 | 22

18. Secondary Outcome: Subject Satisfaction
Description: Subject Satisfaction (Would you have this procedure again?)
Time Frame: 24 months
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 185 | 167 | 39 | 20 | 89
participants
  Definitely Yes | 121 | 86 | 24 | 8 | 62
  Probably Yes | 25 | 32 | 5 | 4 | 9
  Unsure or Too Early to Tell | 10 | 6 | 3 | 2 | 4
  Probably Not | 4 | 3 | 3 | 2 | 3
  Definitely Not | 1 | 2 | 2 | 0 | 0

19. Secondary Outcome: Global Cervical Range of Motion - Change From Baseline
Time Frame: 24 months
Population: As Treated. The difference between the number of treated patients and the number of participants analyzed is due to: death of one randomized ACDF patient, patients who experienced a Device Failure before the 24 month visit, and patients with no data collected for this secondary outcome (missing data).
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Number analyzed (Participants) | 147 | 117 | 35 | 15 | 66
degrees | 5.4 (16.14) | -2.8 (14.67) | 3.0 (14.88) | -14.4 (13.21) | 2.1 (15.36)

20. Secondary Outcome: Average Radiographic Disc Height (mm) - Change From Post-op
Time Frame: 24 months
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate
Number analyzed (Participants) | 153 | 114
mm | -1.0 (0.76) | -1.0 (0.83)

ADVERSE EVENTS:
Time Frame: 24 months. Safety data is still being collected on all DISCOVER subjects through 60 months.
Description: The population used in the adverse event tables is "As Treated". One subject was randomized to control, but was treated with DISCOVER. This explains why the denominators in the adverse event tables are 186 and 166 for the randomized one level cohorts.
Arm/Group | 1-level Cervical TDR | 1-level ACDF With Plate | 2-level Cervical TDR | 2-level ACDF | Training: 1 & 2-level Cervical TDR
Serious Adverse Events (participants affected / at risk) | 59/186 | 44/166 | 14/39 | 5/20 | 24/89
Other Adverse Events (participants affected / at risk) | 158/186 | 135/166 | 38/39 | 20/20 | 83/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-level Cervical TDR (N=186) | 1-level ACDF With Plate (N=166) | 2-level Cervical TDR (N=39) | 2-level ACDF (N=20) | Training: 1 & 2-level Cervical TDR (N=89)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 4 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 3 (4) | 2 (2) | 0 (0) | 3 (3)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Complication of device removal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device migration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dural tear (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Foreign body trauma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture nonunion (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gun shot wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 3 (3)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7) | 1 (1) | 1 (1) | 4 (4)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radicular pain (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal X-ray abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical failure (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Surgical procedure repeated (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thoracic outlet syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulval cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1-level Cervical TDR (N=186) | 1-level ACDF With Plate (N=166) | 2-level Cervical TDR (N=39) | 2-level ACDF (N=20) | Training: 1 & 2-level Cervical TDR (N=89)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Areflexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 9 (9) | 1 (1) | 3 (3) | 4 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 32 (34) | 21 (22) | 7 (7) | 8 (9) | 20 (20)
Bartholin's cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
CSF pressure increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 7 (8) | 5 (6) | 5 (6) | 2 (2) | 5 (5)
Cervical root pain (Nervous system disorders) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 15 (18) | 10 (11) | 3 (4) | 4 (4) | 3 (3)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coeliac disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Contrast media reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis interstitial (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (4)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Device breakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device migration (Injury, poisoning and procedural complications) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Drug intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dural tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 12 (12) | 19 (19) | 8 (8) | 2 (2) | 6 (7)
Dysphasia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Extraskeletal ossification (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Feeling abnormal (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fibrocystic breast disease (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 13 (14) | 5 (7) | 3 (3) | 6 (6)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hoffmann's sign (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Horner's syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 22 (26) | 16 (19) | 12 (18) | 3 (5) | 17 (25)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyporeflexia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incision site oedema (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 6 (6)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (6) | 5 (5) | 2 (3) | 0 (0) | 2 (2)
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hypotension (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Lung hernia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 5 (5) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 4 (4)
Motor dysfunction (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 (20) | 6 (6) | 7 (8) | 1 (1) | 10 (14)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 5 (5) | 6 (6) | 1 (1) | 1 (1) | 2 (2)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 (10) | 4 (5) | 4 (4) | 2 (2) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 4 (4) | 0 (0) | 4 (4)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 54 (71) | 47 (56) | 17 (25) | 9 (9) | 28 (38)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 7 (7) | 3 (3) | 3 (3) | 0 (0) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Myotonia congenita (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 66 (81) | 55 (66) | 24 (38) | 9 (11) | 39 (52)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nerve root compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nerve root lesion (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological symptom (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 41 (50) | 44 (53) | 14 (18) | 8 (17) | 18 (29)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 21 (24) | 13 (17) | 7 (13) | 2 (2) | 10 (15)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Pituitary cyst (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post laminectomy syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (4)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 4 (7) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Purulent discharge (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Radicular pain (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Radicular syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Radiculitis cervical (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiculitis lumbosacral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reflexes abnormal (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 9 (9) | 6 (6) | 2 (2) | 0 (0) | 3 (3)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sensory disturbance (Nervous system disorders) | 1 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal fusion acquired (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stitch abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suture rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thoracic outlet syndrome (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Ulnar neuritis (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paresis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 6 (7)
Vulval cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Whiplash injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment terminated early, and beginning in March 2013, follow-up visits beyond 24 months were limited to Discover subjects only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No